CLINICAL TRIAL: NCT05949463
Title: Effect of an Activity Wristband-based Intermittent Teaching Unit in Physical Education on Students Physical Activity and Its Psychological Mediators: A Cluster-randomized Controlled Trial. School-Fit Study
Brief Title: Activity Wristband-based Intermittent Teaching Unit and Students Physical Activity and Its Psychological Mediators
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valladolid (Other)
Collaborators: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Santiago Guijarro-Romero, Doctor, University of Valladolid
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 1252/CEIH/2020
Record Dates: First submitted 2023-06-30; First posted 2023-07-18 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-07

CONDITIONS: School

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intermittent group (Experimental): The intermittent group students performed an intermittent teaching unit twice a week for eight weeks aimed at promoting healthy physical activity habits. Specifically, the last 15 minutes of each lesson were used. The rest of lessons' time other contents were worked on with no relation to any health physical activity habit (i.e., acrosport, badminton, basketball, volleyball, soccer and athletics).
  Interventions: Other: Intermittent teaching unit
- Control group (Active Comparator): The control group students also carried out two Physical Education lessons a week during the intervention period. During these lessons, contents of handball, basketball, alternative sports and traditional games were developed. However, this group did not wear physical activity activity wristbands or receive any behavior modification specific strategy developed in the intermittent group.
  Interventions: Other: No intervention group

INTERVENTIONS:
Other: Intermittent teaching unit — The intermittent group students performed an intermittent teaching unit twice a week for eight weeks aimed at promoting healthy physical activity habits. Specifically, the last 15 minutes of each lesson were used. The rest of lessons' time other contents were worked on with no relation to any health physical activity habit (i.e., acrosport, badminton, basketball, volleyball, soccer and athletics).
  Arms: Intermittent group
Other: No intervention group — The control group students also carried out two Physical Education lessons a week during the intervention period. During these lessons, contents of handball, basketball, alternative sports and traditional games were developed. However, this group did not wear physical activity activity wristbands or receive any behavior modification specific strategy.
  Arms: Control group

SUMMARY:
Objective: The main objective of the present study was to examine the effects of an intermittent teaching unit based on the use of activity wristbands and behavior modification strategies on high school students perceptions of autonomy support, satisfaction of basic psychological needs, motivation toward Physical Education and physical activity, intention to be physically active, and habitual physical activity levels.

Materials and methods: An initial sample of 353 high school students (final sample = 175; 45.7% females; mean age = 13.3 ± 1.2 years) from two public high schools were cluster-randomly assigned into the intermittent (n = 100) and control (n = 75) groups. The intermittent group performed an intermittent teaching unit twice a week for eight weeks. Specifically, the last 15 minutes of each lesson were used. As the main strategy to promote the practice of regular physical activity, students wore an activity wristband the whole day during the intervention period. Additionally, other behavior modification strategies were also applied (e.g., educational counseling, physical activity goals or reminders). The control group also performed two Physical Education sessions a week during the intervention period, but without using wristbands or other behavior modification strategies. Before and after the intervention, as well as at the end of the follow-up period (six weeks), students' physical activity practice mediators and physical activity levels were measured by validated questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Being enrolled in the seventh to tenth grade at the secondary education level
* Participating in the normal Physical Education lessons
* Being exempt of any health problem that would make them unable to engage in physical activity normally
* Presenting the corresponding signed written consent by their legal tutors
* Presenting their own corresponding signed written assent

Exclusion Criterion:

- Not having performed the evaluation of the dependent variables correctly at the pre-intervention, post-intervention and/or follow-up measures following the administration rules (being removed only for incomplete variables and not for the overall study)

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 175 (Actual)
Dates: Start 2022-01-10 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Change in Perceived autonomy support | Pre-intervention, immediately post-intervention, and after 6-week follow-up
  The Physical Education teacher autonomy-support was assessed through the Spanish version of the Multi-Dimensional Perceived Autonomy Support Scale for Physical Education (MD-PASS-PA). It consists of 15 items (five items per factor) that assessed organizational, procedural, and cognitive autonomy support. The items were preceded by the statement "My Physical Education teacher...". The Spanish version of MD-PASS-PA has shown adequate psychometric properties among adolescents.
Change in Basic psychological needs | Pre-intervention, immediately post-intervention, and after 6-week follow-up
  Students' perceptions of autonomy, competence, and relatedness satisfaction in Physical Education and physical exercise were assessed using the Spanish version of the Basic Psychological Needs in Exercise Scale (BPNES). It consists of 12 items (four items per factor) that assessed autonomy, competence and relatedness. The items were preceded by the statement "When I do physical activity…". The Spanish version of BPNES has shown adequate psychometric properties among adolescents.
Change in Motivation toward Physical Education | Pre-intervention, immediately post-intervention, and after 6-week follow-up
  Participants' self-determined motivation toward Physical Education was measured by the Spanish version of the Revised Perceived Locus of Causality Scale (PLOC-R). It consists of of 23 items spread over six dimensions (four items each except external regulation) that measure intrinsic motivation, amotivation, integrated, identified, introjected, and external regulation. This questionnaire was preceded by the statement "I participate in Physical Education lessons…". The autonomous (i.e., averaging intrinsic, integrated, and identified regulation) and controlled (i.e., averaging introjected and external) motivations were also calculated. The Spanish version of the PLOC-R has shown adequate psychometric properties among adolescents.
Change in Self-determined motivation towards physical activity | Pre-intervention, immediately post-intervention, and after 6-week follow-up
  Students' motivation towards physical activity was measured using the Spanish version of the Behavioral Regulation in Exercise Questionnaire (BREQ-3). It consists of 23 items distributed into six dimensions (four items each except identified regulation) that measure intrinsic motivation, amotivation, integrated, identified, introjected, and external regulation. This questionnaire was preceded by the statement: "I do physical activity...". The autonomous and controlled motivations were also calculated. The Spanish version of the BREQ-3 has shown adequate psychometric properties among high-school students.
Change in Intention to be physically active | Pre-intervention, immediately post-intervention, and after 6-week follow-up
  Students' intention to be physically active in their free time was measured using the Spanish version of the Intention to partake in leisure-time physical activity questionnaire. It is composed of three items. The items were preceded by the sentence: "In my free time, after school ...". The Spanish version of this questionnaire has shown adequate psychometric properties among adolescents.
Change in Habitual physical activity | Pre-intervention, immediately post-intervention, and after 6-week follow-up
  Students' habitual physical activity was measured using the Physician-based Assessment and Counseling for Exercise questionnaire (PACE). It consists of two questions that measure how many days in the last week and in a habitual week at least 60 minutes of physical activity are performed. A 7-point Likert-type scale, ranging from 0 to 7 was used. The PACE questionnaire has shown adequate psychometric properties among high-school students.

CONTACTS AND LOCATIONS:
Locations (1):
- Santiago Guijarro-Romero, Valladolid, Spain

REFERENCES:
- [Derived] Guijarro-Romero S, Mayorga-Vega D, Casado-Robles C, Viciana J. Effect of an activity wristband-based intermittent teaching unit in Physical Education on students' physical activity and its psychological mediators: a cluster-randomized controlled trial. School-fit study. Front Psychol. 2023 Sep 20;14:1228925. doi: 10.3389/fpsyg.2023.1228925. eCollection 2023. PMID 37799526